CLINICAL TRIAL: NCT00099892
Title: Efficacy and Safety of Vildagliptin in Combination With Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2303
Record Dates: First submitted 2004-12-21; First posted 2004-12-22 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: vildagliptin

SUMMARY:
Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. The purpose of this study is to assess the safety and effectiveness of two doses of vildagliptin, an unapproved drug, when added to metformin in people with type 2 diabetes who are not at target blood glucose levels on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Blood glucose criteria must be met
* On a stable dose of metformin as defined by the protocol
* Body mass index (BMI) in the range 22-45

Exclusion Criteria:

* Type 1 diabetes
* Pregnancy or lactation
* Evidence of serious diabetic complications
* Evidence of serious cardiovascular complications
* Laboratory value abnormalities as defined by the protocol
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 544 (Actual)
Dates: Start 2004-05; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c after 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose at 24 weeks
Patients with endpoint HbA1c <7% after 24 weeks
Patients with reduction in HbA1c >/=to 0.7% after 24 weeks
Change from baseline in body weight at 24 weeks
Change from baseline in fasting lipids at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Bosi E, Camisasca RP, Collober C, Rochotte E, Garber AJ. Effects of vildagliptin on glucose control over 24 weeks in patients with type 2 diabetes inadequately controlled with metformin. Diabetes Care. 2007 Apr;30(4):890-5. doi: 10.2337/dc06-1732. Epub 2007 Feb 2. PMID 17277036